CLINICAL TRIAL: NCT04285320
Title: Intravesical Antibiotic Instillations Versus Oral Suppression for the Treatment of Recurrent Urinary Tract Infections in Post-menopausal Women
Brief Title: Antibiotic Bladder Instillations vs. Oral Suppression for the Treatment of Recurrent Urinary Tract Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, charbel salamon, Director, Urogynecology Division & Fellowship, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1565199
Record Dates: First submitted 2020-02-17; First posted 2020-02-26 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: Antibiotic bladder instillation; Intravesical antibiotic instillation; Oral suppressive therapy; Recurrent UTI
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravesical antibiotic instillation (Active Comparator)
  Interventions: Drug: Intravesical antibiotic instillation
- Oral antibiotic suppressive therapy (Active Comparator)
  Interventions: Drug: Antibiotic oral suppressive therapy

INTERVENTIONS:
Drug: Intravesical antibiotic instillation — Based on the participant's allergy and antibiotic resistance profile, one of the following three antibiotics will be instilled intravesically via a latex free BARD® 12 French Foley catheter for a total of 6-8 instillations (2 instillations/week) according to the Atlantic Health System Urogynecology Division antibiotic bladder instillation standard protocol:
  * Amikacin-30 mg in 60 ml of sterile water
  * Gentamycin-80mg in 60ml sterile water
  * Tobramycin-80 mg in 100 ml of sterile water
  Arms: Intravesical antibiotic instillation
Drug: Antibiotic oral suppressive therapy — In the antibiotic oral suppression therapy arm, one of the following routinely used antibiotics will be prescribed for a total of 3 months according to the American Urogynecology Society Guidelines and based on the participant's allergy and antibiotic resistance profile:
  * Trimethoprim daily (100 mg)
  * Trimethoprim/sulfamethoxazole daily (40 mg/200 mg)
  * Trimethoprim/sulfamethoxazole every 3 days (40 mg/200 mg)
  * Nitrofurantoin monohydrate/macrocrystals daily (50 mg)
  * Nitrofurantoin monohydrate/macrocrystals daily (100 mg)
  * Cephalexin daily (125 mg)
  * Cephalexin daily (250 mg)
  * Fosfomycin every 10 days (3 grams)
  Arms: Oral antibiotic suppressive therapy

SUMMARY:
This is a research study that aims to determine if antibiotic bladder instillations (placing an antibiotic directly into the bladder) over several sessions at the office is a good option to prevent recurrent urinary tract infections, in comparison with oral suppression therapy (taking daily antibiotics in the form of pills by mouth). Oral antibiotic suppression therapy is currently the most common treatment route for recurrent urinary tract infections in post-menopausal women. The bladder antibiotic instillation may overcome the disadvantages of oral suppression therapy such as antibiotic resistance, certain side effects, and recurrence of infections after finishing the treatment course.

DETAILED DESCRIPTION:
In this study, the investigators aim to determine the effectiveness of intra-vesical antibiotic instillations for the prophylactic treatment of recurrent urinary tract infections in menopausal women in comparison with oral suppressive therapy. This is a parallel un-blinded randomized-controlled trial. the investigators will randomize post-menopausal women with recurrent urinary tract infections to either receive 6-8 intra-vesical antibiotic instillations at the office or to receive 3 months of oral antibiotic suppressive therapy.

In the bladder instillation arm, based on the participant's allergy and antibiotic resistance profile, one of the following three antibiotics will be instilled intravesically via a latex free BARD® 12 French Foley catheter for a total of 6-8 instillations (2 instillations/week) according to the Atlantic Health System Urogynecology Division antibiotic bladder instillation standard protocol:

* Amikacin-30 mg in 60 ml of sterile water
* Gentamycin-80mg in 60ml sterile water
* Tobramycin-80 mg in 100 ml of sterile water

In the antibiotic oral suppression therapy arm, one of the following routinely used antibiotics will be prescribed for a total of 3 months according to the American Urogynecology Society Guidelines and based on the participant's allergy and antibiotic resistance profile:

* Trimethoprim daily (100 mg)
* Trimethoprim/sulfamethoxazole daily (40 mg/200 mg)
* Trimethoprim/sulfamethoxazole every 3 days (40 mg/200 mg)
* Nitrofurantoin monohydrate/macrocrystals daily (50 mg)
* Nitrofurantoin monohydrate/macrocrystals daily (100 mg)
* Cephalexin daily (125 mg)
* Cephalexin daily (250 mg)
* Fosfomycin every 10 days (3 grams) All medications used in this study are approved by the FDA to treat urinary tract infections.

Participants will be followed for total of 3 months after finishing either treatment course by only reviewing their medical records to collect data regarding development of urinary tract infections after treatment.

Primary endpoint/outcome:

• To compare the number of women developing urinary tract infections during the 3 months following treatment between the two groups.

Secondary endpoints/outcomes:

* To compare the rate of antibiotic resistance of isolated pathogens after intravesical antibiotic instillation vs. oral antibiotic suppressive therapy
* To compare side effects of the two treatment modalities

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women with recurrent urinary tract infections (2 infections in a 6-month period or at least 3 infections in a 1-year period)
* Receiving estrogen vaginal therapy for 1 month prior to enrollment
* Able to come in to the office twice weekly for 3-4 weeks
* English speaking
* No allergy to at least one of the three antibiotics used for bladder instillations and at least one of the four antibiotics recommended for oral suppressive therapy.
* No uro-pathogen resistance to at least one of the three antibiotics used for bladder instillations and at least one of the four antibiotics recommended for oral suppressive therapy.

Exclusion Criteria:

* Allergy to all study antibiotics (Gentamicin, Tobramycin, Amikacin, Trimethoprim/sulfamethoxazole, Fosfomycin, Nitrofurantoin and Cephalexin)
* Recent Urine culture with pathogens resistant to all study antibiotics (Gentamicin, Tobramycin, Amikacin, Trimethoprim/sulfamethoxazole, Fosfomycin, Nitrofurantoin and Cephalexin)
* Renal failure (Creatinine clearance <30ml/min)
* History of urinary retention
* History of genitourinary structural abnormalities

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants with urinary tract infections following treatment course | Assessed starting immediately after the treatment is completed for a total of 3 months.
  To compare the percentage of women developing urinary tract infections during the 3 months following treatment between the two groups.

SECONDARY OUTCOMES:
The rate of antibiotic resistance of pathogens in participants developing urinary tract infections after completing the treatment course. | Assessed starting immediately after the treatment is completed for a total of 3 months
  To compare the rate of antibiotic resistance of isolated pathogens when participants develop a urinary tract infection during the 3 months follow up period after intra-vesical antibiotic instillation vs. oral antibiotic suppressive therapy. the percentage of antibiotics on the susceptibility list of urine cultures will be compared between participants developing urinary tract infection in each group during the 3 months follow-up period after completing the treatment.
the percentage of patients developing side effects of the 2 treatments | From the date of randomization until the date of first documented side effect assessed up to 3 months after the treatment is completed in each arm
  To compare the percentage of patients developing side effects between the two treatment modalities. At their routine follow up visits patients will be asked about whether or not they developed side effects and the type and severity of side effects of the treatment received. The percentage of patients developing side effects (per type and severity) in each arm will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Charbel Salamon, MD, MS, Principal Investigator — Atlantic Health System - Morristown Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chernyak S, Salamon C. Intravesical Antibiotic Administration in the Treatment of Recurrent Urinary Tract Infections: Promising Results From a Case Series. Female Pelvic Med Reconstr Surg. 2020 Feb;26(2):152-154. doi: 10.1097/SPV.0000000000000810. PMID 31990805